CLINICAL TRIAL: NCT03103464
Title: Sit-to-Stand Progression Using Movi Chair vs Traditional Practices
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No one consented for this study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lavon Beard, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X161207007
Record Dates: First submitted 2017-03-28; First posted 2017-04-06 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Patient's primary physical therapist will not be aware whether the patient is in the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Patients to receive standard-of-care physical therapy + sit-to-stand therapy using the Movi chair 3x/wk.
  Interventions: Other: Standard-of-Care Therapy + Sit-to-Stand Therapy
- Control Group (Active Comparator): Patients to receive standard-of-care physical therapy 3x/wk.
  Interventions: Other: Standard-of-Care Therapy

INTERVENTIONS:
Other: Standard-of-Care Therapy + Sit-to-Stand Therapy — Standard-of-care physical therapy 3x/wk for approximately 30 minutes each time + sit-to-stand training using the Movi chair 3x/wk for approximately 10 minutes each time.
  Arms: Intervention Group
Other: Standard-of-Care Therapy — Standard-of-care physical therapy 3x/wk for approximately 30 minutes each time.
  Arms: Control Group

SUMMARY:
Prior to discharging admitted patients, current UAB Hospital policy recommends physical therapy intervention for patients with impaired functional mobility. However, UAB Hospital currently does not have a standardized physical therapy protocol to rehabilitate admitted patients with impaired functional mobility who require moderate assist (defined as physical therapist expending 25-50% effort to assist the patient in standing). In order to reduce the effect of impaired mobility, numerous interventions have been employed at UAB. As a result, there is great variability of treatment procedures performed by various physical therapists to help moderate assist patients return to their level of functioning prior to hospital admission. The purpose of the study is three-fold: 1) to evaluate whether a proposed physical therapy protocol using a commercially available medical device, the Movi chair, contributes to improved mobility for moderate assist patients, 2) to investigate how patient rate of rehabilitation to prior level of functioning is similar/different with the proposed physical therapy protocol using Movi vs the current non-standardized practice for moderate assist patients, and 3) to compare patient confidence in physical therapy with Movi vs the current non-standardized practice using survey for moderate assist patients. In addition, we will track participant's disposition i.e. continued motor and functional change following discharge from the hospital through review of physical therapy records.

DETAILED DESCRIPTION:
Most activities of daily living require unassisted ability to stand from a sitting position. Therefore, physical therapy exercises aimed at improving this essential action are critically important for patients with impaired functional mobility. Although sit-to-stand tests are a well-known tool used to assess physical function, they have only recently has been proposed for systematic strength training.

Those patients who would most benefit from sit-to-stand training require moderate assist or greater. However, these patients have significant difficulty initiating sit-to-stand exercises from a horizontal chair surface and have been largely excluded from prior studies examining sit-to-stand for strength training. These patients have been excluded not only because they cannot safely stand on their own, but also because manually lifting these patients poses a significant lifting-injury risk to physical therapists.

Movi is a commercially available hybrid mechanical lift and chair who's key feature is a built in battery powered motor (rated for 600 lbs) that pivots on its axis to raise and lower a patient up to 20 degrees. We believe that this feature represents an opportunity for introducing sit-to-stand strength training to previously excluded moderate assist patients. Progressively lowering the chair's angle of inclination over consecutive physical therapy sessions will allow the patient to practice sit-to-stand at a reduced effort until the to horizontal angle is reached.

As sit-to-stand strength training is a concept only proposed in 2011, no previous studies exist concerning a sit-to-stand physical therapy protocol using a chair progressively lowering the seat's angle of inclination. Currently, therapists use their clinical judgment when approaching patients with difficulty standing by utilizing exercise, skill repetition, in addition to other strengthening strategies and equipment to reach goals. Timed sit-to-stand has already been used at UAB in order to test a patient's progress in physical therapy but not as a therapy protocol in itself, partly because equipment allowing progressive lowering of the seat's angle of inclination has not been available until now. This study was conceived due to the great variability of physical therapy in the Hospital setting and the critical need for standardization and evaluating a protocol that has potential to positively impact patient speed and ease of recovery to prior level of functioning.

The therapy protocol utilizing the Movi chair will include the following:

1. Mobilize patient to Movi chair (via lift or manual transfer)
2. Document lowest height in 5 degree increments (in degrees from inclinometer attached to Movi chair) where patient is able to complete a sit-to-stand transfer with minimal assistance (defined as requiring < 25% effort from the physical therapist) allowing patient to use his or her arms on thighs or armrests if needed.
3. The patient will perform 5 sit-to-stand transfers from this level, rest until recovery, and do additional sets to increase muscle strength only if able.
4. During subsequent visits, patient will begin at prior set level. If able to perform a sit-to-stand transfer with less than minimal assistance, the elevation of the chair will be lowered by 5 degree increments until able to complete a sit-to-stand transfer with minimal assistance or greater and the patient will perform sit-to-stand transfer repetitions from the new height.
5. This protocol will continue until the patient is able to perform a sit-to-stand transfer from a standard height chair with supervision assistance or until the patient is discharged to the next level of care

i. Once able to complete a sit-to-stand transfer from a standard height, a five-time-sit-to-stand (FTSST) will be performed 3 times per week.

Treatment of the control group will utilize standard recliners and traditional therapy methods (transfer training, therapeutic exercise). Once an investigator consents the patient for the study, if the patient has been randomized to either control group or intervention group, a non-investigator physical therapist will perform his or her usual physical therapy exercises to minimize bias from study investigators completing therapy. Investigators will test FTSST time for patients in the control group 3 times per week. Only investigators will treat the intervention group using the above outlined protocol 3 times per week. Once intervention group patients are able to complete a sit-to-stand transfer from a standard height, a FTSST will be performed 3 times per week by a study investigator. Investigators will also record the Hierarchical Assessment of Balance and Mobility (HABAM) score for intervention group patients when they test FTSST time as an added measure of mobility. The HABAM is an interval level mobility instrument that is already in use as a valid and reliable mobility instrument in the older acute medical population. This score does not require any additional exercises with the patient beyond the FTSST. Investigators will ask the non-investigator physical therapists caring for the control group patients to estimate control group patients' HABAM, which can be easily estimated after working with the patient during routine standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving physical therapy at UAB hospital that require moderate assistance or greater with sit-to-stand transfers during initial evaluation
* Patients with baseline function of supervision as obtained in the initial physical therapy (PT) evaluation
* Patients who have an inpatient hospital stay of at least 4 days

Exclusion Criteria:

* Patients with diagnoses that are progressive in nature
* Patients in intensive care units due to critical medical condition and confounding factors
* Patients with cognitive impairment as noted in the medical record
* Patients with weight bearing precautions other than free weight bearing (FWB) or weight bearing as tolerated (WBAT)
* Children (under the age of 18), prisoners and pregnant women
* Patients who are not able to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Rate of progression from moderate to minimal assist | Through study completion, an average of 2 weeks
  Patient rate of progression from moderate (<50% assistance from physical therapist) to minimal (<25% assistance from physical therapist) assist during hospital admission

SECONDARY OUTCOMES:
Hierarchical Assessment of Balance and Mobility Score | Through study completion, an average of 2 weeks
  Score grading the patient on balance, mobility, and transfers on a 0-28 scale
Five-time sit-to-stand time | Through study completion, an average of 2 weeks
  Time for patient to complete sit-to-stand 5x from standard chair

CONTACTS AND LOCATIONS:
Overall Officials: Lavon Beard, DPT, MBA, Principal Investigator — Manager Physical Therapy, Doctor of Physical Therapy
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No